CLINICAL TRIAL: NCT01345994
Title: Brain Plasticity in Carpal Tunnel Syndrome and Its Response to Acupuncture
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martinos Center for Biomedical Imaging (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Vitaly Napadow, Massachusetts General Hospital
Other Study IDs: AT004714; R01AT004714-01 (NIH)
Record Dates: First submitted 2011-04-25; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture - local (Experimental): acupuncture on forearm only
  Interventions: Procedure: electro-acupuncture
- acupuncture - distal (Experimental): acupuncture on both arm and leg
  Interventions: Procedure: electro-acupuncture

INTERVENTIONS:
Procedure: electro-acupuncture — acupuncture stimulation with electricity

SUMMARY:
This study will characterize brain plasticity in Carpal Tunnel Syndrome and will determine how this central fMRI biomarker is modulated by acupuncture. This study will also investigate the behavioral consequences of maladaptive cortical plasticity in this disease population.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 20-60.
2. History

   * Pain and/or paresthesia in median nerve distribution (i.e., numbness in some combination of digit 1, 2, 3, and the radial part of digit 4)
   * Nocturnal pain and/or paresthesia in median nerve distribution
   * Symptoms (a and b) greater than 3 months in duration
3. Physical Exam with two of the following three findings:

   * Phalen's and Durkin's sign (positive with paresthesia in at least 1 of 3 radial digits)
   * Abnormal grip strength (greater than 2 S.D. compared to uninvolved side using an isometric hand grip device)
4. Nerve conduction findings consistent with mild to severe CTS:

Mild CTS: Delayed distal latency of the sensory nerve conductions across the wrist (> 3.7milliseconds and/or > than 0.5 milliseconds compared to the ulnar sensory conduction) with normal motor conductions

Moderate CTS: Delayed distal latency of the sensory nerve conductions across the wrist as stated above with delayed distal latency of the motor conductions across the wrist (> 4.2 milliseconds).

Severe CTS: Delayed distal latency of the sensory nerve conductions across the wrist as stated above with greater than 50% loss of motor amplitudes (relative to unaffected side and/or normative range).

Exclusion Criteria:

1. Contraindications to MRI examination (pregnancy, pacemaker, etc. according to guidelines set by MGH NMR-Center)
2. History of diabetes mellitus or other major cardiovascular, respiratory, or neurological illnesses.
3. History of rheumatoid arthritis.
4. History of wrist fracture with direct trauma to median nerve.
5. Current usage of prescriptive opioid pain medication.
6. Severe thenar atrophy.
7. Nerve entrapment other than median nerve.
8. Cervical radiculopathy or myelopathy.
9. Generalized peripheral neuropathy.
10. A blood dyscrasia or coagulopathy or current use of anticoagulation therapy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2009-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Functional MRI brain response | Baseline vs. Post-Acupuncture (average 9 weeks later)
  Several fMRI outcomes will be assessed including brain hyperactivity and somatotopy

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States